CLINICAL TRIAL: NCT01006876
Title: Role of Coumadin in Preventing Periprocedural Thrombo-Embolism as a Complication of Radio Frequency Catheter Ablation in High-risk Atrial Fibrillation Patients
Brief Title: Role of Coumadin in Preventing Thromboembolism in Atrial Fibrillation (AF) Patients Undergoing Catheter Ablation
Acronym: COMPARE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Texas Cardiac Arrhythmia Research Foundation (Other)
Collaborators: University of Kansas (Other); California Pacific Medical Center (Other); Stanford University (Other); Case Western Reserve University (Other); Southlake Regional Health Centre (Other); Catholic University, Italy (Other)
Responsible Party: Principal Investigator, Andrea Natale, Medical director, Texas Cardiac Arrhythmia Research Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TCAI-COMPARE
Record Dates: First submitted 2009-11-02; First posted 2009-11-03 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Thromboembolism
Keywords: coumadin; peri-procedural thromboembolism; RFCA; high risk atrial fibrillation
MeSH Terms: conditions — Thromboembolism | interventions — Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study Arm (Active Comparator): Patients receive continuous Coumadin therapy throughout the study.
  Interventions: Drug: Coumadin
- Control Arm (Active Comparator): Patients discontinue Coumadin 3-4 days prior to ablation and replace it with heparin until the end of the procedure and bridge low molecular weight heparin (LMWH) with Coumadin 48-72 hours after ablation.
  Interventions: Drug: Coumadin

INTERVENTIONS:
Drug: Coumadin — Continuous oral Coumadin therapy through the catheter ablation procedure
  Other Names: warfarin
  Arms: Study Arm
Drug: Coumadin — Patients discontinue Coumadin 3-4 days prior to ablation and replace it with heparin until the end of the procedure and bridge low molecular weight heparin (LMWH) with Coumadin 48-72 hours after ablation.
  Other Names: Warfarin
  Arms: Control Arm
Drug: Coumadin — Oral tablets, daily dose, till the therapeutic INR of 2-3 is achieved
  Other Names: Warfarin

SUMMARY:
This study aims to explore the risk of periprocedural thromboembolic events in continuous versus interrupted Coumadin therapy in a large, randomized high-risk patient population undergoing radio-frequency catheter ablation for atrial fibrillation.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common arrhythmia encountered in clinical practice, affecting 2.3 million people in the United States (1). A major cause of stroke, AF substantially increases the risk of thromboembolism which necessitates oral anticoagulation therapy (OAT) for high-risk patients. Radiofrequency percutaneous catheter ablation (RFCA) is an effective strategy for the treatment of symptomatic drug-refractory atrial fibrillation. However, periprocedural cerebrovascular accident (CVA) due to thrombus or air embolism remains one of the most serious complications of AF ablation. In spite of precautions taken before, during, and after the ablation to minimize the risk of CVA, the reported event rate remains 0.5-2.8% (2).

The incidence of thromboembolic events is dependent on the extensiveness of the ablation procedure as well as the periprocedural anticoagulation strategy (2). Some studies have described charring and soft thrombus formation when the temperature exceeds 100 degree C during RFCA, which probably is caused by blood protein denaturation and coagulation (3). Currently an open saline irrigation-tip ablation catheter (3.5 mm Thermocool catheter) is used which reduces the thermal injury by keeping the temperature under control (4), while enabling the operator to use high wattage RF energy to effectively ablate the arrhythmogenic focus.

The two most utilized periprocedural OAT strategies are; 1) discontinuation of Coumadin three to five days prior to ablation, utilization of heparin or enoxaparin before the procedures, and "bridging" low molecular weight heparin with Coumadin after ablation, and 2) RFCA with continuation of Coumadin before, during and after the procedure (2) without any change in dosage. Limited data are available regarding the risk of thromboembolism with and without periprocedural Coumadin in AF patients undergoing catheter ablation .The aim of this prospective randomized study is to evaluate the effect of the above two OAT strategies on the incidence of TE within 48 hours post-RFCA.

Patient Selection, Treatment and Follow-up Period:

Patients randomized as study group would continue Coumadin without any periprocedural change while undergoing catheter ablation. Those randomized as control group would discontinue Coumadin 3-4 days prior to ablation and replace it with heparin till the end of the procedure and bridge LMWH with Coumadin 48-72 hours after ablation.

An INR of 2-3 would be ascertained in all patients prior to procedure. Patients with subtherapeutic INR would not be included in this study.

Procedure: Coumadin therapy would be started at least two months prior to the ablation in order to achieve the therapeutic INR at least three weeks prior to the procedure.

Anticoagulation strategy I (Coumadin interrupted): Twice daily until the evening prior to ablation procedure, 0.5-1 mg/kg of enoxaparin would be administered and bridged to Coumadin. At the time of the procedure, enoxaparin would be replaced by heparin. At the end of the procedure, the sheaths would be removed during full anticoagulation. After the procedure heparin would be discontinued, and protamine 10 to 15 mg would be given. Sheaths would be pulled when activated clotting time (ACT) would be <250 seconds. Aspirin 325 mg would be given before the patient leaves the electrophysiology laboratory. Warfarin would be administered the evening of pulmonary vein isolation. Enoxaparin 1 mg/kg BID and 0.5 mg/kg BID would be routinely started and would be stopped when the INR is > 2. Patients with LSPAF, left ventricular dysfunction or history of thrombo-embolism would receive overlapping anticoagulation with enoxaparin for three days after the procedure. The remaining patients would receive a double dose of Coumadin on the night of the ablation followed by the routine pre-procedure dose from the next day.

Anticoagulation strategy II (continuous Coumadin): Coumadin would not be discontinued in this group of patients. The INR would be monitored every week for four weeks preceding the ablation and it should be above 2.0. All patients in AF on the day of the procedure where an INR above 2 is not demonstrable for four consecutive weeks preceding the procedure would undergo TEE.

PVAI would be done while on Coumadin treatment. No heparin or enoxaparin would be administered to any patient prior to the procedure. Before transseptal punctures, a heparin bolus (100 to 150 U/Kg) would be administered to all patients. During the procedure, the infusion rate would be adjusted to keep the activated clotting time in the range of 350 to 450 sec.

After the procedures, heparin infusion would be stopped and anticoagulation would be reversed with 10 to 15 mg of Protamine, and sheaths would be pulled when the activated clotting time is less than 250 sec. Patients would receive 325 mg of Aspirin before leaving the EP lab. They would continue their Coumadin dosage regimens with no changes before or after the procedure aiming to an INR of 2 to 3.

Following randomization, patients are considered to be in the treatment period 2 months before the procedure to 48-72 hours after the procedure.

Ablation Procedure: Standard radiofrequency catheter ablation procedure based on physician's discretion would be followed.

All patients will undergo baseline and post-procedure MRI within 24-hours of the procedure.

Follow-up period is 48 hours post-procedure; during which all patients would have neurologic evaluation; at the end of the procedure and every four hours for the next 48 hours. Clinical neurologic evaluation would include assessment of mental status such as ability to pay attention, memory, judgment and orientation to self, place and time; maneuvers to test the cranial nerves, assessment of motor functions by testing strength in different muscle groups and assessment of sensory functions by evaluating touch, pain, vibration and positional awareness as well as the deep tendon reflexes.

Patients with questionable neurologic impairment would undergo neuroimaging evaluations like head CT or MRI.

ELIGIBILITY:
Inclusion Criteria:

1. Age- 18-75 years
2. Patients in paroxysmal, persistent or long-standing persistent (LSP) AF
3. patients with CHADS2 score ≥ 1
4. AF patients with INR in the range of 2.0-3.0 in the last 3-4 weeks prior to ablation

Exclusion Criteria:

1. Patients with known bleeding disorders or inherited thrombophilic disorder
2. Patients with oral contraceptives or estrogen replacement therapy
3. Patients with prosthetic heart valves
4. Patients unable or willing to give informed consent
5. Contraindications for Coumadin therapy
6. Patients with CHADS2 score zero
7. Contraindication to undergoing an MRI

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1584 (Actual)
Dates: Start 2010-01; Primary Completion 2013-03 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Absence of thromboembolic events 48 hours post-ablation | 48 hours

SECONDARY OUTCOMES:
Recurrence of AF and late thromboembolic events | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Natale, MD, Principal Investigator — Texas Cardiac Arrhythmia Institiute
Locations (1):
- St.David's Medical Center, Austin, Texas, United States

REFERENCES:
- [Derived] Bawazeer GA, Alkofide HA, Alsharafi AA, Babakr NO, Altorkistani AM, Kashour TS, Miligkos M, AlFaleh KM, Al-Ansary LA. Interrupted versus uninterrupted anticoagulation therapy for catheter ablation in adults with arrhythmias. Cochrane Database Syst Rev. 2021 Oct 21;10(10):CD013504. doi: 10.1002/14651858.CD013504.pub2. PMID 34674223
- [Derived] Di Biase L, Burkhardt JD, Santangeli P, Mohanty P, Sanchez JE, Horton R, Gallinghouse GJ, Themistoclakis S, Rossillo A, Lakkireddy D, Reddy M, Hao S, Hongo R, Beheiry S, Zagrodzky J, Rong B, Mohanty S, Elayi CS, Forleo G, Pelargonio G, Narducci ML, Dello Russo A, Casella M, Fassini G, Tondo C, Schweikert RA, Natale A. Periprocedural stroke and bleeding complications in patients undergoing catheter ablation of atrial fibrillation with different anticoagulation management: results from the Role of Coumadin in Preventing Thromboembolism in Atrial Fibrillation (AF) Patients Undergoing Catheter Ablation (COMPARE) randomized trial. Circulation. 2014 Jun 24;129(25):2638-44. doi: 10.1161/CIRCULATIONAHA.113.006426. Epub 2014 Apr 17. PMID 24744272